CLINICAL TRIAL: NCT05830045
Title: A Study Evaluates the Safety, Pharmacokinetics, Immunogenicity and Efficacy of QLP2117 in Advanced Solid Tumor Patients
Brief Title: A Phase I Study of QLP2117 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLP2117-101
Record Dates: First submitted 2023-04-04; First posted 2023-04-26 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ia： QLP2117 Dose escalation and PK expansion (Experimental)
  Interventions: Drug: QLP2117
- Ib：QLP2117 Dose expansion (Experimental)
  Interventions: Drug: QLP2117

INTERVENTIONS:
Drug: QLP2117 — Specified dose on specified days

SUMMARY:
This is the first in human study of QLP2117. To evaluate the Safety, Pharmacokinetics, Immunogenicity and Efficacy of QLP2117 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmation of recurrent or refractory advanced solid tumours, and have progressed on standard therapy, or are intolerable for available standard therapy, or there is no available standard therapy.
2. At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1(phase Ia dose escalation only requires at least one assessable lesion)
3. Eastern Cooperative Oncology Group Performance Status of 0 or 1
4. Agree to provide archived tumor tissue samples of primary or metastatic lesions.
5. Have adequate organ function as described in the protocol.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding
2. HBsAg/HBcAb positive and HBV-DNA>1000 copy/mL;HCV-Ab positive and detection of HCV-RNA suggested viral replication
3. Is currently participating and receiving study medication in another study within 4 week prior to the first dose of study treatment
4. Has an active autoimmune disease that has required systemic treatment in past 2 years.
5. Has an active infection requiring systemic therapy
6. Has received a live vaccine wihtin 30 days of planned start of study treatment
7. Has know history of, or any evidence of interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | 21days
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | up to 96 weeks
Objective Response Rate for phase 1b | up to 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Ruihua, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No